CLINICAL TRIAL: NCT03687216
Title: A Single-center Randomized Controlled Study of Secondary Prophylaxis of Cirrhosis Related Esophagogastric Variceal Hemorrhage Treated With HVPG-guided Therapy or Standard Esophageal Variceal Ligation Plus Beta-blocker
Brief Title: HVPG-Guided Therapy Versus EVL Plus NSBB in Second Prophylaxis of Esophageal Variceal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Director of Department of Gastroenterology and Hepatology, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HGT-EN
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Esophageal Varices in Cirrhosis of the Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVPG group (Experimental): HVPG-guided therapy (TIPS or EVL plus NSBB according to HVPG)
  Interventions: Procedure: HVPG-guided therapy
- Routing group (Active Comparator): Routing therapy (EVL plus NSBB)
  Interventions: Procedure: Routing Therapy

INTERVENTIONS:
Procedure: HVPG-guided therapy — The baseline HVPG measurement is performed. According to the result, patients with an HVPG over 20 mmHg will be receive transjugular intrahepatic portocaval shunt (TIPS) .
  Patients with an HVPG below 20 mmHg will be treated by endoscopic variceal ligation (EVL) plus nonselective beta blocker (NSBB) propranolol until treatment fails.
  Arms: HVPG group
Procedure: Routing Therapy — Without HVPG measurement, patients receive endoscopic variceal ligation (EVL) plus nonselective beta blocker (NSBB) propranolol.
  Arms: Routing group

SUMMARY:
A single-center randomized controlled study comparing endoscopic or interventional therapy guided by the hepatic venous pressure gradient (HVPG) , to standard endosopic variceal ligation plus nonselective beta-blocker therapy (NSBB) in patients with esophageal varices due to liver cirrhosis with a history of esophageal variceal hemorrhage.Primary study outcome of the study is variceal rebleeding episodes occurring within the first years after interventions. Second study outcomes of the study are hepatic encephalopathy occurrence, mortality occurrence, liver transplantation or other cirrhosis-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosed by clinical examination, imaging or biopsy;
* A previous history of variceal hemorrhage;
* Written informed consent.

Exclusion Criteria:

* Previous history of secondary prophylactic treatment;
* Contraindications to treatment of endoscopy, surgery and TIPS
* Severe cardiac, pulmonary or renal dysfunction;
* Lactating or pregnant;
* Malignancies;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Variceal rebleeding rate | One year of follow-up
  The incidence of clinically significant gastrointestinal variceal bleeding

SECONDARY OUTCOMES:
Hepatic encephalopathy: The incidence of hepatic encephalopathy | One year of follow-up
  The incidence of hepatic encephalopathy
Ascites: The incidence of ascites detected by ultrasound | One year of follow-up
  The incidence of ascites detected by ultrasound
Cirrhotic complications | One year of follow-up
  portal vein thrombosis, liver dysfunction, hepatorenal syndrome et al.
Liver transplant-free survivial | One year of follow-up
  Time from the procedure to the date of lost-to-follow-up or death or liver transplant

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No